CLINICAL TRIAL: NCT02156804
Title: A Single-Arm, Open-Label, Multicenter Clinical Trial With Nivolumab (BMS-936558) for Subjects With Histologically Confirmed Stage III (Unresectable) or Stage IV Melanoma Progressing Post Prior Treatment Containing an Anti-CTLA4 Monoclonal Antibody
Brief Title: A Single-Arm, Open-Label, Multicenter Clinical Trial With Nivolumab (BMS-936558) for Subjects With Histologically Confirmed Stage III (Unresectable) or Stage IV Melanoma Progressing Post Prior Treatment Containing an Anti-CTLA4 Monoclonal Antibody (CheckMate 172)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-172; 2014-001286-28 (EudraCT Number)
Record Dates: First submitted 2014-05-29; First posted 2014-06-05 (Estimated); Results first posted 2020-02-20 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab (BMS-936558) (Experimental): Nivolumab (BMS-936558) Intravenous solution every 2 weeks
  Interventions: Drug: Nivolumab (BMS-936558)

INTERVENTIONS:
Drug: Nivolumab (BMS-936558)

SUMMARY:
The purpose of this study is to determine the rate and frequency of high-grade (CTCAE v4.0 Grade 3 or higher), treatment-related, select adverse events in subjects with histologically confirmed stage III (unresectable) or stage IV melanoma and progression post prior treatment containing an anti-Cytotoxic T Lymphocyte Antigen (CTLA-4) monoclonal antibody, treated with Nivolumab (BMS-936558) at a dose of 3 mg/kg every two weeks.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with histologically confirmed malignant melanoma
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS):

  * PS 0 to 1
  * PS 2
* Previously treated unresectable stage III or stage IV melanoma as per the American Joint Committee on Cancer 2010 Guidelines regardless of BRAF mutation status
* Subjects must have experienced evaluable Response Evaluation Criteria In Solid Tumors (RECIST 1.1)-defined disease progression
* Prior treatment with chemotherapy, interferon (adjuvant setting), Interleukin (IL-2), BRAF/MEK inhibitors for subjects with known BRAF mutations, Mitogen-activated or extracellular signal- regulated protein kinase (MEK) inhibitors for Neuroblastoma Ras Viral (v-ras) oncogene homolog (NRAS) mutations, and cKIT inhibitor subjects with known cKIT mutations are allowed
* Patients with CNS metastases are eligible:

  * if CNS metastases are treated, patients are asymptomatic or neurologically returned to baseline
  * if they have previously untreated CNS metastases and are asymptomatic
  * if they have leptomeningeal metastases, are treated and asymptomatic or neurologically returned to baseline with life expectancy > 3 months
* Patients with a known history of Grades 3-4 immune-related adverse reactions during/after anti-CTLA-4 therapy if all toxicities have resolved at least to Grade 1

Exclusion Criteria:

* Subjects with untreated, active Central Nervous System (CNS) metastases are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1009 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (152):
- Austria (6):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Salzburg
  - Local Institution, Sankt Pölten
  - Local Institution, Vienna
  - Local Institution, Wein
- Belgium (9):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Local Institution, Edegem
  - Local Institution, Ghent
  - Local Institution, Hasselt
  - Az Groeninge, Kortrijk
  - Local Institution, Leuven
  - Chu De Liege, Liège
- Czechia (3):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- Finland (4):
  - Local Institution, Helsinki
  - Local Institution, Jyväskylä
  - Local Institution, Oulu
  - Local Institution, Tampere
- Germany (39):
  - Local Institution, Lübeck, Schleswig-Holstein
  - Local Institution, Augsburg
  - Local Institution, Bochum
  - Local Institution, Buxtehude
  - Local Institution, Chemnitz
  - Local Institution, Cologne
  - Local Institution, Dessau
  - Local Institution, Dresden
  - Local Institution, Erfurt
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Gera
  - Local Institution, Giessen
  - Local Institution, Göttingen
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Heilbronn
  - Local Institution, Jena
  - Local Institution, Kassel
  - Local Institution, Kiel
  - Local Institution, Leipzig
  - Local Institution, Ludwigshafen
  - Local Institution, Magdeburg
  - Local Institution, Mainz
  - Local Institution, Marburg
  - Local Institution, Minden
  - Local Institution, München
  - Local Institution, Münster
  - Local Institution, Nuremberg
  - Local Institution, Quedlinburg
  - Local Institution, Recklinghausen
  - Local Institution, Regensburg
  - Local Institution, Schwerin
  - Local Institution, Traunstein
  - Local Institution, Tübingen
  - Local Institution, Wurzbug
- Greece (3):
  - Local Institution, Heraklion, Crete
  - Local Institution, Athens
  - Local Institution, Thessaloniki
- Hungary (5):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Pécs
  - Local Institution, Szeged
  - Local Institution, Szombathely
- Ireland (4):
  - Local Institution, Wilton, CORK
  - Local Institution, Dublin
  - Local Institution, Galway
  - Local Institution, Waterford
- Italy (12):
  - Local Institution, Bari
  - Local Institution, Bergamo
  - Local Institution, Genova
  - Local Institution, Meldola (FC)
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Palermo
  - Local Institution, Roma
  - Local Institution, Siena
  - Local Institution, Terni
  - Local Institution, Torino
- Local Institution, Luxembourg, Luxembourg
- Netherlands (14):
  - Local Institution, Amsterdam, North Holland
  - Local Institution, Amsterdam
  - Local Institution, Breda
  - Local Institution, Enschede
  - Local Institution, Groningen
  - Local Institution, Leeuwarden
  - Local Institution, Leiden
  - Local Institution, Maastrict
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
  - Local Institution, Sittard-Geleen
  - Local Institution, Utrecht
  - Local Institution, Veldhoven
  - Local Institution, Zwolle
- Norway (3):
  - Local Institution, Ålesund
  - Local Institution, Bergen
  - Local Institution, Oslo
- Poland (4):
  - Local Institution, Bydgoszcz
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Warsaw
- Portugal (2):
  - Local Institution, Lisbon
  - Local Institution, Porto
- Romania (2):
  - Local Institution, Bucharest
  - Local Institution, Romania
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Spain (16):
  - Local Institution, Albacete
  - Local Institution, Barcelona
  - Local Institution, Bilbao
  - Local Institution, Donostia / San Sebastian
  - Local Institution, Granada
  - Local Institution, Las Palmas de Gran Canaria
  - Local Institution, Madrid
  - Hospital De Madrid, Norte Sanchinarro, Madrid
  - Local Institution, Málaga
  - Local Institution, Oviedo
  - Local Institution, Palma de Mallorca
  - Local Institution, Salamanca
  - Hospital Clinico Univ. de Santiago-CHUS, Santiago de Compostela
  - Local Institution, Seville
  - Local Institution, Toledo
  - Local Institution, Valencia
- Sweden (2):
  - Local Institution, Lund
  - Local Institution, Uppsala
- Switzerland (5):
  - Local Institution, Aarau
  - Local Institution, Basel
  - Local Institution, Bellinzona
  - Local Institution, Chur
  - Local Institution, Zurich
- United Kingdom (16):
  - Local Institution, Bristol, AVON
  - Local Institution, Northwood, Middlesex
  - Local Institution, Birmingham
  - Local Institution, Cambridge
  - Local Institution, Cottingham
  - Local Institution, Essex
  - Local Institution, Glasgow
  - Local Institution, London
  - Local Institution, Manchester
  - Local Institution, Metropolitan Borough of Wirral
  - Local Institution, Newcastle upon Tyne
  - Local Institution, Oxford
  - Local Institution, Southampton
  - Local Institution, Surrey
  - Local Institution, Swansea
  - Local Institution, Truro

REFERENCES:
- [Derived] Schadendorf D, Ascierto PA, Haanen J, Espinosa E, Demidov L, Garbe C, Guida M, Lorigan P, Chiarion-Sileni V, Gogas H, Maio M, Fierro MT, Hoeller C, Terheyden P, Gutzmer R, Guren TK, Bafaloukos D, Rutkowski P, Plummer R, Waterston A, Kaatz M, Mandala M, Marquez-Rodas I, Munoz-Couselo E, Dummer R, Grigoryeva E, Young TC, Nathan P. Safety and efficacy of nivolumab in challenging subgroups with advanced melanoma who progressed on or after ipilimumab treatment: A single-arm, open-label, phase II study (CheckMate 172). Eur J Cancer. 2019 Nov;121:144-153. doi: 10.1016/j.ejca.2019.08.014. Epub 2019 Sep 30. PMID 31581055
- [Derived] Nathan P, Ascierto PA, Haanen J, Espinosa E, Demidov L, Garbe C, Guida M, Lorigan P, Chiarion-Sileni V, Gogas H, Maio M, Fierro MT, Hoeller C, Terheyden P, Gutzmer R, Guren TK, Bafaloukos D, Rutkowski P, Plummer R, Waterston A, Kaatz M, Mandala M, Marquez-Rodas I, Munoz-Couselo E, Dummer R, Grigoryeva E, Young TC, Schadendorf D. Safety and efficacy of nivolumab in patients with rare melanoma subtypes who progressed on or after ipilimumab treatment: a single-arm, open-label, phase II study (CheckMate 172). Eur J Cancer. 2019 Sep;119:168-178. doi: 10.1016/j.ejca.2019.07.010. Epub 2019 Aug 21. PMID 31445199
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1009 participants were enrolled into the study , 1008 wrere treated, 1 participants was not treated due to withdrew consent
Groups:
- Nivolumab 3mg/kg: Nivolumab 3 mg/kg as a 60-minute IV infusion every 2 weeks
Period: Overall Study
Arm/Group | Nivolumab 3mg/kg
Started | 1009
Completed | 1008
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Arm/Group | Nivolumab 3mg/kg
Number analyzed (Participants) | 1008
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 451
  Male | 557
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 972
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 987
  More than one race | 0
  Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: the Incidence of Highgrade (CTCAE v4.0 Grade 3 or Higher), Treatment Related,Select Adverse Events.
Description: The number of participants who reported high-grade (CTCAE v4.0 Grade 3 or higher), treatment-related, select AEs (pulmonary,gastrointestinal, skin, renal, hepatic, endocrine) were summarized using the all treated analysis set by system organ class and Medical Dictionary for Regulatory (MedDRA) preferred term.
Time Frame: Up to 2 years
Population: All treated participants
Measure: Number; unit: Number of Participants
Arm/Group | Nivolumab 3mg/kg
Number analyzed (Participants) | 1008
Number of Participants
  Gastrointestinal Adverse events (Grade 3-4) | 16
  Gastrointestinal adverse events (Grade 5) | 0
  Hepatic adverse events (Grade 3-4) | 30
  Hepatic adverse events (Grade 5) | 0
  Pulmonary adverse events(Grade 3-4) | 6
  Pulmonary adverse events(Grade 5) | 0
  Renal adverse events (Grade 3-4) | 4
  Renal adverse events (Grade 5) | 0
  Skin adverse events ( Grade 3-4) | 13
  Skin adverse events ( Grade 5) | 0
  Hypersensitivity adverse event( Grade 3-4) | 1
  Hypersensitivity adverse event( Grade 5) | 0
  Endocrine adverse events(Grade 3-4) | 18
  Endocrine adverse events(Grade 5) | 0

2. Secondary Outcome: The Incidence of All High-grade (Grades 3 and Higher), Select Adverse Events
Description: The number of Participants who reported high-grade (CTCAE v4.0 Grade 3 or higher), select AEs were summarized using the all treated analysis set by system organ class and MedDRA preferred term.
Time Frame: Up to 2 years
Population: All treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Nivolumab 3mg/kg
Number analyzed (Participants) | 1008
Number of Participants
  Gastrointestinal Adverse events (Grade 3-4) | 24
  Gastrointestinal adverse events (Grade 5) | 0
  Hepatic adverse events (Grade 3-4) | 52
  Hepatic adverse events (Grade 5) | 1
  Pulmonary adverse events(Grade 3-4) | 7
  Pulmonary adverse events(Grade 5) | 1
  Renal adverse events (Grade 3-4) | 12
  Renal adverse events (Grade 5) | 1
  Skin adverse events ( Grade 3-4) | 19
  Skin adverse events ( Grade 5) | 0
  Hypersensitivity adverse event( Grade 3-4) | 2
  Hypersensitivity adverse event( Grade 5) | 0
  Endocrine adverse events(Grade 3-4) | 24
  Endocrine adverse events(Grade 5) | 0

3. Secondary Outcome: Median Time to Onset (Grades 3-4) of Select Adverse Events
Description: Select AEs were summarized according to their incidence as well as their time to onset.
Time Frame: Up to 2 years.
Population: All Treated Participants.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Nivolumab 3mg/kg
Number analyzed (Participants) | 1008
Weeks
  Endocrine Adverse Events | 12 [0.3 to 88.4]
  Gastrointestinal Adverse Events | 23.50 [0.3 to 93.0]
  Hepatic Adverse Events | 10.14 [0.1 to 116.0]
  Pulmonary Adverse Events | 14.86 [1.3 to 64.9]
  Renal Adverse Events | 11.71 [1.1 to 60.0]
  Skin Adverse Events | 34.36 [1.1 to 88.0]
  Hypersensitivity/infusion reaction Adverse Events | 29.57 [29.57 to 29.57]

4. Secondary Outcome: Median Time to Resolution (Grades 3-4) of Select Adverse Events
Description: Select AEs were summarized according to their incidence as well as their time to resolution
Time Frame: Up to 2 years
Population: All Treated Participants
Measure: Median (Full Range); unit: Weeks
Arm/Group | Nivolumab 3mg/kg
Number analyzed (Participants) | 1008
Weeks
  Endocrine Adverse Events | 2.43 [0.4 to 138.0]
  Gastrointestinal Adverse Events | 3.71 [0.1 to 85.9]
  Hepatic Adverse Events | 9.43 [0.1 to 128.1]
  Pulmonary Adverse Events | 2.57 [0.1 to 20.4]
  Renal Adverse Events | 1.93 [1.29 to 3.29]
  Skin Adverse Events | 5.07 [0.1 to 121.1]
  Hypersensitivity/infusion reaction Adverse Events | 0.29 [0.29 to 0.29]

5. Secondary Outcome: Overall Survival
Description: The time from first dosing date to the date of death.
Time Frame: Up to 4 years
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab 3mg/kg
Number analyzed (Participants) | 1008
Months | 21.2 [18.2 to 24.4]

ADVERSE EVENTS:
Time Frame: Between first dose and 30 days after last dose ( up to 2 years)
Groups:
- NIVOLUMAB 3 MG/KG IV: Nivolumab 3 mg/kg as a 60-minute IV infusion every 2 weeks
Arm/Group | NIVOLUMAB 3 MG/KG IV
All-Cause Mortality (participants affected / at risk) | 527/1008
Serious Adverse Events (participants affected / at risk) | 593/1008
Other Adverse Events (participants affected / at risk) | 857/1008
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 3 MG/KG IV (N=1008)
Anaemia (Blood and lymphatic system disorders) | 10
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocarditis (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Addison's disease (Endocrine disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 5
Autoimmune thyroiditis (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 4
Hypopituitarism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 3
Lymphocytic hypophysitis (Endocrine disorders) | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 1
Steroid withdrawal syndrome (Endocrine disorders) | 1
Ectropion (Eye disorders) | 1
Iridocyclitis (Eye disorders) | 1
Iritis (Eye disorders) | 1
Macular hole (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 13
Ascites (Gastrointestinal disorders) | 5
Autoimmune colitis (Gastrointestinal disorders) | 3
Autoimmune pancreatitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 7
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 14
Dyspepsia (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Ileal perforation (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal fistula (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 4
Intussusception (Gastrointestinal disorders) | 2
Large intestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 5
Chest pain (General disorders) | 2
Disease progression (General disorders) | 2
Fatigue (General disorders) | 7
General physical health deterioration (General disorders) | 22
Generalised oedema (General disorders) | 1
Malaise (General disorders) | 3
Nodule (General disorders) | 1
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 9
Sudden death (General disorders) | 3
Treatment failure (General disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 8
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 3
Hepatomegaly (Hepatobiliary disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 4
Jaundice (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Contrast media allergy (Immune system disorders) | 2
Drug hypersensitivity (Immune system disorders) | 1
Abdominal infection (Infections and infestations) | 4
Abdominal sepsis (Infections and infestations) | 2
Anal abscess (Infections and infestations) | 1
Appendiceal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 6
Conjunctivitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 3
Device related sepsis (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 7
Escherichia urinary tract infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Haematoma infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infected dermal cyst (Infections and infestations) | 1
Infected lymphocele (Infections and infestations) | 1
Infection (Infections and infestations) | 5
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 9
Lung infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 13
Pneumonia legionella (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 5
Sepsis (Infections and infestations) | 8
Septic encephalopathy (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 11
Urosepsis (Infections and infestations) | 4
Vascular device infection (Infections and infestations) | 1
Viral diarrhoea (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Dose calculation error (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 5
Procedural headache (Injury, poisoning and procedural complications) | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
CSF test abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
General physical condition abnormal (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Lipase increased (Investigations) | 2
Pancreatic enzymes increased (Investigations) | 1
Transaminases increased (Investigations) | 2
Troponin T increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Fistula (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 278
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Altered state of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 3
Brachial plexopathy (Nervous system disorders) | 2
Brain injury (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 3
Brain stem haemorrhage (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 7
Encephalopathy (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 3
Facial paralysis (Nervous system disorders) | 2
Facial paresis (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Hemiparesis (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Hypertensive encephalopathy (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Miller Fisher syndrome (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Narcolepsy (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 3
Peripheral nerve lesion (Nervous system disorders) | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 6
Sensorimotor disorder (Nervous system disorders) | 2
Spinal cord compression (Nervous system disorders) | 4
Status epilepticus (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Device dislocation (Product Issues) | 1
Confusional state (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Personality change (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 9
Autoimmune nephritis (Renal and urinary disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Postrenal failure (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 2
Ureteric stenosis (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 2
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Penile oedema (Reproductive system and breast disorders) | 1
Testicular oedema (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 3
Angiopathy (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 4
Jugular vein thrombosis (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 3
Peripheral venous disease (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Vascular occlusion (Vascular disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery insufficiency (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Adrenal haemorrhage (Endocrine disorders) | 1
Retinal detachment (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Anal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Pain (General disorders) | 1
Gastroenteritis viral (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Psychotic disorder (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Lymphocele (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVOLUMAB 3 MG/KG IV (N=1008)
Anaemia (Blood and lymphatic system disorders) | 126
Hypothyroidism (Endocrine disorders) | 114
Abdominal pain (Gastrointestinal disorders) | 102
Abdominal pain upper (Gastrointestinal disorders) | 58
Constipation (Gastrointestinal disorders) | 132
Diarrhoea (Gastrointestinal disorders) | 210
Nausea (Gastrointestinal disorders) | 212
Vomiting (Gastrointestinal disorders) | 120
Asthenia (General disorders) | 168
Fatigue (General disorders) | 295
Oedema peripheral (General disorders) | 81
Pyrexia (General disorders) | 130
Nasopharyngitis (Infections and infestations) | 88
Urinary tract infection (Infections and infestations) | 54
Alanine aminotransferase increased (Investigations) | 83
Aspartate aminotransferase increased (Investigations) | 78
Blood alkaline phosphatase increased (Investigations) | 52
Lipase increased (Investigations) | 79
Weight decreased (Investigations) | 63
Decreased appetite (Metabolism and nutrition disorders) | 143
Arthralgia (Musculoskeletal and connective tissue disorders) | 148
Back pain (Musculoskeletal and connective tissue disorders) | 116
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 55
Myalgia (Musculoskeletal and connective tissue disorders) | 62
Pain in extremity (Musculoskeletal and connective tissue disorders) | 93
Headache (Nervous system disorders) | 122
Insomnia (Psychiatric disorders) | 55
Cough (Respiratory, thoracic and mediastinal disorders) | 134
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 81
Dry skin (Skin and subcutaneous tissue disorders) | 54
Pruritus (Skin and subcutaneous tissue disorders) | 115
Pruritus generalised (Skin and subcutaneous tissue disorders) | 89
Rash (Skin and subcutaneous tissue disorders) | 54
Vitiligo (Skin and subcutaneous tissue disorders) | 77
Dry mouth (Gastrointestinal disorders) | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT02156804/SAP_000.pdf
  • Study Protocol (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT02156804/Prot_001.pdf